CLINICAL TRIAL: NCT04971655
Title: The Effect of Music Therapy on Anxiety and Pain in Individuals With Type 2 Diabetes Who Just Started Insulin Therapy
Brief Title: The Effect of Music Therapy on Pain and Anxiety
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Satı Can, Principal Investigator, Abant Izzet Baysal University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: AIBU-SBF-SC-01
Record Dates: First submitted 2021-06-22; First posted 2021-07-21 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: diabetes; insulin; pain; anxiety; music therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Insulin Resistance; Pain; Anxiety Disorders | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: two groups with a music therapy group and control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music therapy group (Experimental): When individuals with diabetes apply to diabetes education after their polyclinic examination, music therapy will be applied in addition to routine monitoring and applications throughout the education. Turkish Folk, Classical, Turkish Art and Sufi Music genres will be offered as options to the individuals in the intervention group and will be listened to throughout the process. During the training, the selected music will be played over the loudspeaker. Before the training, this group; Patient Description Form and Spielberger State-Trait Anxiety Scale will be applied. After the training, Visual Analogue Scale and State Anxiety Scale will be applied.
  Interventions: Other: Music therapy
- Control group (No Intervention): When individuals apply to diabetes education after their polyclinic examinations, routine monitoring and application will be made throughout the education. Before the training, this group; Patient Description Form and Spielberger State-Trait Anxiety Scale will be applied. After the training, Visual Analogue Scale and State Anxiety Scale will be applied.

INTERVENTIONS:
Other: Music therapy — Music therapy will be applied throughout diabetes education. Turkish Folk, Classical, Turkish Art and Sufi Music genres will be offered to individuals as an option and will be listened to throughout the process. Instrumental works will be uploaded to the computer by the researchers and will be played on the loudspeaker during the training.
  Arms: Music therapy group

SUMMARY:
The effect of music therapy on pain and anxiety will be evaluated in individuals with diabetes who start insulin therapy for the first time. Music will be played during the training.

DETAILED DESCRIPTION:
The prevalence of diabetes is increasing all over the world. Prevention of diabetes complications by providing glycemic control is the most important goal of diabetes treatment. Timely initiation of insulin therapy may be advantageous in ensuring glycemic control. Insulin therapy should be started without delay, especially in patients with Type 2 diabetes, in cases such as other diseases that intervene and increase the need for insulin, severe insulin resistance, surgery, pregnancy or progression of diabetes complications. However, most people with diabetes are reluctant to start insulin therapy, which may delay the start of treatment. In particular, he is reluctant to start insulin therapy for reasons such as the thought that insulin will limit his life, the concern that insulin is harmful, the expectation of pain due to injection, the worry that he will not be able to make insulin successfully, the fear of hypoglycemia, and that he will have to use insulin constantly. This situation can cause negative diabetes outcomes such as poor glycemic, diabetes complications, increased risk of death and disability. For this reason, sufficient time should be taken to address insulin-related concerns and persuaded to use insulin. In studies, music therapy is used as a supportive care intervention, as a noninvasive nursing intervention, music therapy is used to reduce pain and anxiety and increase compliance. Music, which is called the food of the soul, has been used by many civilizations in the treatment of physiological and psychological problems since ancient times. The use of music for therapeutic purposes since ancient civilizations has led to the emergence of the concept of music therapy. Music therapy has shown serious developments in the historical process, especially at the end of the 20th century. Experimentally, music therapy has been used, and it has been observed that scientific studies have been carried out to improve the physical and psychological conditions of the patients, especially during and after the procedure. As a result of the studies, it has been shown that music has positive effects on human health, affects human activities and has positive cognitive effects. However, the effect of conditions such as the type of music and the preference of the patient is also in question in achieving this effect. For this reason, it is important to determine the type of music specific to the person and the disease in terms of positive effect.

When the literature is examined, it is seen that music therapy is used in different areas such as mental health, diabetic foot ulcer management, neuropathic pain, glucose control in individuals with diabetes and positive results are obtained. This study was planned as a randomized controlled study to determine the effect of insulin injection on reducing pain and anxiety in diabetic individuals who were started on insulin therapy for the first time.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and over
* Able to speak and understand Turkish
* No hearing problem
* With place and time orientation
* Does not have any psychiatric disease
* Insulin therapy for the first time
* Volunteers will be included in the study

Exclusion Criteria:

* Under 18 years old
* Does not speak Turkish
* Hearing problems
* No place and time orientation
* Having any psychiatric disease
* Non-volunteer individuals will not be included in the study

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2021-08-04 (Actual); Primary Completion 2022-06-28 (Estimated); Study Completion 2022-07-15 (Estimated)

PRIMARY OUTCOMES:
Visual Pain Scale (VAS) | one hours
  The patient assigns a value between 0 and 10 for pain. On the scale, there is '0' no pain, '10' very severe pain levels. The patient marks his current state on this line. The length of the distance from the point where there is no pain to the point marked by the patient gives the pain score. 1-4 points: mild pain, 5-6 points: moderate pain, 7 points and above: severe pain.
State-Trait Anxiety Inventory (STAI) | one hours
  The scale consists of two parts:
  1. State Anxiety Scale: It is a 4-point Likert-type scale consisting of 20 questions aiming to measure how individuals feel themselves at the moment. The scores obtained from the scale range from 20 to 80, with high scores indicating high anxiety and low scores indicating low anxiety levels. 0-19 points from the scale indicate that there is no anxiety, 20-39 points indicate mild, 40-59 points moderate, 60-79 points indicate the level of severe anxiety, and a score above 60 indicates the need for professional help.
  2. Trait Anxiety Scale: It indicates how the person feels during the process, regardless of the situation and conditions. The scores obtained from the scale vary between 20 and 80, and a high score indicates a high level of anxiety, and a low score indicates a low level of anxiety. 0-30 indicates low anxiety, 31-49 indicates moderate anxiety, and 50 and higher indicates high anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Saadet CAN ÇİÇEK, Ph.D, Study Director — Bolu Abant Izzet Baysal University, Health Sciences Faculty, Department of Nursing
Locations (1):
- SATI CAN, Bolu, Merkez, Turkey (Türkiye)